CLINICAL TRIAL: NCT01618539
Title: A Prospective Study to Establish a Correlation Between Infusion Rate of Propofol and Bispectral Index (BIS) in Patients Receiving Total Intravenous Anesthesia (TIVA)
Brief Title: Correlation of Bispectral Index Score and Total Intravenous Anesthesia (TIVA)
Status: Terminated | Type: Observational
Why Stopped: PI retired prior to final N number reached
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 2011001109
Record Dates: First submitted 2012-06-05; First posted 2012-06-13 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2016-07

CONDITIONS: Benign/Malignant Neoplasm; Long Bone Fracture
Keywords: Total intravenous anesthesia, Bispectral Index Score
MeSH Terms: conditions — Neoplasms | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: propofol — varying intravenous dosages

SUMMARY:
General Anesthesia is usually produced by an intravenous agent and then maintained with a breathing agent till the surgery is completed. However, there is a recent trend to produce and maintain general anesthesia solely with an intravenous agent, such as propofol, in view of its advantages. This delivery method is called Total Intravenous Anesthesia (TIVA). The depth of general anesthesia can be measured by an anesthetic depth monitoring device called Bispectral Index (BIS). The use of BIS to determine the depth of anesthesia has been well established whenever a breathing agent is used to maintain general anesthesia. However, the validity of using BIS with TIVA has not been adequately investigated. This study will compare the BIS values at different doses of TIVA in order to establish any correlation between the two. If such a correlation is established, BIS monitoring can safely be recommended to determine anesthetic depth under TIVA.

DETAILED DESCRIPTION:
Pre-anesthetic Management: This research will be initiated after receiving an approval from the Institution Review Board, and an informed written consent will be obtained from each patient. Forty patients in the age range 18-65 years and presenting for elective orthopedic or gynecological procedures will be recruited. Both male and female patients will be considered. Only patients with American Society of Anesthesiologists (ASA) physical status I, II and III will be included. Patients who are pregnant and those with uncontrolled hypertension with BP above 180/100, unstable angina, chronic obstructive lung disease requiring oxygen therapy at home, and end-stage liver and kidney diseases will be excluded. In addition, orthopedic surgery that needs the patient in prone position will not be eligible for this investigation. Patients who have a medication allergy to propofol and food allergy to egg and soy, since egg lecithin and soy milk are constituents of propofol preparation, will be excluded. In order to have a complete data collection, only surgical procedures scheduled to last more than three hours will be considered for this study.

Anesthetic Management: Routine anesthetic care, such as intravenous line placement and American Society of Anesthesiologists' standard monitoring, will be applied to all patients. In addition, a non-invasive Bispectral Index (BIS) sensor will be placed on patient's forehead and connected to its monitor. Midazolam (25mcg/kg) and fentanyl (1mcg/kg) will be administered to establish preanesthetic sedation and analgesia, respectively. Lidocaine 40mg will be given to attenuate propofol-induced injection pain. Thereafter, Total Intravenous Anesthesia (TIVA) will be induced with propofol (2mg/kg), and tracheal intubation facilitated with a neuromuscular blocking agent chosen by the attending anesthesiologist. The skeletal muscle relaxation will be maintained as needed for the surgical procedure. The TIVA will be maintained with propofol infusion, for approximately half-hour, at 160mcg/kg/min with minor adjustment, as needed, to maintain patient's vital signs within ± 20% of the baseline. Once a steady state is established, propofol infusion rate will be reduced to 140mcg/kg/min and maintained for approximately 15-30 min, following which the infusion rate will be increased to 180mcg/kg/min and maintained for the same period of time. Thereafter, the propofol infusion rate will be returned to 160mcg/kg/min. This exercise will be repeated at 120mcg/kg/min and 200mcg/kg/min if patient's vital signs permit. In addition, remifentanil at an infusion rate of 0.02 - 0.2mcg/kg/min will be administered to provide surgical analgesia during the general anesthetic period. The infusion rate of remifentanil will be tailored to the demands of the surgical stimulation. During the study period, the attending anesthesiologist will have the option to deviate from the study protocol and adjust the propofol infusion rate, as needed, to maintain patient's vital signs within ± 20% of the baseline if such a need arises. An independent observer will continuously monitor the BIS values at all time frames. Following the study period needed to collect the required data, the attending anesthesiologist will have the option to continue general anesthesia with either TIVA or with the traditional inhalational anesthetic. The reversal of the neuromuscular blockade and subsequent tracheal extubation, at the conclusion of surgery, will be performed using the customary criteria employed in anesthetic practice. In addition, the routine protocols used for surgical infection prevention and attenuation of postoperative pain and vomiting will be followed.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 undergoing orthopedic or gyn surgery
* ASA status I-III

Exclusion Criteria:

* pregnant patients
* uncontrolled hypertension with B/P above 180/100
* unstable angina
* end stage liver or kidney disease
* Pts anticipated to be placed in prone position for surgery
* Documented allergy to propofol, eggs, soy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
BIS response to varying TIVA dosages | 3 hours
  Correlation between various infusion rates of propofol administered during TIVA and BIS values during the first 3 hours of the operative procedure

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shulman, MD, Principal Investigator — Rutgers/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No